CLINICAL TRIAL: NCT00646711
Title: A 14 Day Randomized, Open-Label, Cross-Over, Single Center, Outpatient Study of Depakote Delayed-Release or Depakote Sprinkle vs. Divalproex Sodium Extended-Release in Child and Adolescent Patients With Epilepsy
Brief Title: Pediatric Switch Study for Children and Adolescent Patients With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sharon Stec, Assoc Director, Abbott
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M02-461
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Pediatric Epilepsy
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence Group I (Experimental): Depakote Delayed Release/Depakote Sprinkle
  Interventions: Drug: Depakote Delayed-Release/Depakote Sprinkle
- Sequence Group II (Experimental): Depakote ER
  Interventions: Drug: Depakote ER

INTERVENTIONS:
Drug: Depakote Delayed-Release/Depakote Sprinkle — Administered according to the subject's usual regimen.
  Other Names: ABT-711; Depakote DR; Depakote Sprinkle; divalproex sodium
  Arms: Sequence Group I
Drug: Depakote ER — Dose converted to 8-20% higher than Depakote DR or Depakote Sprinkle.
  Other Names: ABT-711; Depakote Extended Release; divalproex sodium
  Arms: Sequence Group II

SUMMARY:
To assess the tolerability of switching from Depakote Sprinkle Capsules or Depakote tablets to Depakote ER tablets in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with a clinical diagnosis of epilepsy considered stable by the investigator.
* Must be in good physical health, on the same dose of all medications, including Depakote and other AEDs, for 2 week period prior to randomization.
* Minimum body weight of 37 lbs.

Exclusion Criteria:

* Six-month history of drug or alcohol abuse.
* Status epilepticus within 6 months prior to screening.
* Abnormal platelet or ALT/AST levels.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2003-02; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Number of seizures | 2 weeks
Number of Adverse Events | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond, Virginia, United States